CLINICAL TRIAL: NCT00004431
Title: Randomized Study of L-Baclofen in Patients With Refractory Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13391; UPSOM-950686-9608; UPSOM-FDR000914
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-04

CONDITIONS: Trigeminal Neuralgia
Keywords: neurologic and psychiatric disorders; rare disease; trigeminal neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia; Neurologic Manifestations; Mental Disorders; Rare Diseases

INTERVENTIONS:
Drug: L-baclofen

SUMMARY:
OBJECTIVES: I. Evaluate the efficacy of L-baclofen in patients with refractory trigeminal neuralgia.

II. Evaluate the safety and tolerance of L-baclofen in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, parallel study.

Patients are randomized to receive either L-baclofen or placebo orally at increasing daily doses for 1 week. Patients then continue to receive the maximum dosage acceptable for a 1 week maintenance period.

Patients, thereafter, may enroll in a long term open label study with L-baclofen.

Patients are followed at 1, 3, 6, 9, and 12 months.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Idiopathic trigeminal neuralgia - Paroxysmal attacks of facial or frontal pain lasting a few seconds to less than 2 minutes - Pain has at least 4 of the following characteristics: Distribution along one or more divisions of the trigeminal nerve Sudden, intense, sharp, superficial, stabbing, or burning quality Pain intensity severe Precipitation from trigger areas, or by certain daily activities such as eating, talking, washing the face, or cleaning the teeth Between paroxysms entirely asymptomatic - No neurological deficit - Attacks are stereotyped in the individual patient - Exclusion of other causes of facial pain by history, physical examination and special investigations when necessary Must be uncontrolled or refractory as defined by occurrence of at least 2 paroxysms of pain per day despite conventional treatment with maximally tolerated doses of carbamazepine --Prior/Concurrent Therapy-- No concurrent medication for trigeminal neuralgia other than carbamazepine, phenytoin, and neurontin Concurrent medication for other conditions allowed Concurrent medication must be on stable dose(s) --Patient Characteristics-- Hepatic: No significant hepatic disease Renal: No significant renal disease Neurological: No evidence of progressing neurological disorder (e.g., intracranial neoplasm, multiple sclerosis) Other: No history of drug abuse Not pregnant Effective contraception required of all fertile patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-06; Study Completion 1999-09

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Soso, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States